CLINICAL TRIAL: NCT06222450
Title: Rock Steady: A Mobile, Gamified Vestibular Rehabilitation Therapy App for Adults With Dizziness Related to Mild Traumatic Brain Injury
Brief Title: Vestibular Rehabilitation App for Adults With Dizziness Related to mTBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mountain Home Research & Education Corporation (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TP210512
Record Dates: First submitted 2024-01-16; First posted 2024-01-24 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Mild Traumatic Brain Injury; Dizziness
Keywords: vestibular rehabilitation; digital health; remote therapeutic monitoring
MeSH Terms: conditions — Brain Concussion; Dizziness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard VRT (Active Comparator): The gaze stabilization, habituation and balance/gait HEP will be delivered using standard paper handouts
  Interventions: Behavioral: Vestibular Rehabilitation Therapy (VRT)
- Digital VRT (Experimental): The gaze stabilization, habituation and balance/gait HEP will be delivered using a digital home program using the Health in Motion platform
  Interventions: Behavioral: Vestibular Rehabilitation Therapy (VRT)

INTERVENTIONS:
Behavioral: Vestibular Rehabilitation Therapy (VRT) — customized VRT home exercise program per standard of care, includes gaze stabilization, habituation, balance and gait exercises, and endurance training

SUMMARY:
The goal of this clinical trial is to compare outcomes for standard vestibular rehabilitation home program to a digital vestibular rehabilitation home program in adults with dizziness related to mild traumatic brain injury (mTBI). The main question is whether participants who use the digital format of vestibular rehabilitation improve to a greater extent at discharge than those who use the standard format. Participants will undergo a customized vestibular rehabilitation home exercise program per standard of care, consisting of gaze stabilization, habituation, balance and gait exercises, and endurance training under the supervision of a physical therapist. Participants will complete the gaze stabilization and habituation exercises 2-3 times per day and the balance and gait exercises 1 time per day for 4 weeks.

Participants will be tested before and after the 4-week intervention. At the initial session, the researcher will perform standard clinical tests of the inner ear balance system. Also at the initial session, the researcher will perform standard clinical tests of balance and walking and questionnaires about the impact of dizziness on daily activities. At the final session, the researcher will repeat the tests of balance and walking and questionnaires. Three months after completing the intervention participants will complete an online questionnaire about the impact of dizziness on daily activities.

DETAILED DESCRIPTION:
A single blind randomized controlled trial (RCT) will be performed with pre- and post-treatment assessment and a 3-month follow-up assessment. Study groups are defined by the method that the home exercise vestibular rehabilitation therapy (VRT) program is provided: Group 1 will receive standard vestibular rehabilitation therapy (S-VRT) home program, while Group 2 will receive a digital vestibular rehabilitation therapy (D-VRT) home program using the Health in Motion platform. Sixty-eight adults (+10% for attrition) with sub-acute (2 weeks-3 months) or chronic dizziness (> 3 months) related to mTBI will be recruited and enrolled in the study. We will use a randomized block design to assure equal allocation of symptom severity to the intervention groups. Random assignment will be made using SPSS random number function. The research coordinator at each study site will create sealed study envelopes with the random study identification number that contains group assignment. In order to instruct the participant in the appropriate exercise intervention, the treating physical therapist will receive an envelope (in consecutive order) once a subject has consented to participate in the study. This study will incorporate a single blind research design, so that the researcher performing clinical balance and gait assessments will be blinded to group assignment. It is not possible to blind the treating therapist or participants.

During the pre-test session, the researcher will perform a standard vestibular evaluation including tests of balance and walking as well as questionnaires about dizziness impact on activities, balance confidence, motion sensitivity, and disability.

The treating clinician will create and provide a customized VRT home exercise program (HEP) per standard of care, consisting of gaze stabilization, habituation, balance and gait exercises, and endurance training. Gaze stabilization exercises involve head movement while maintaining fixation on a target which may be stationary or moving. Habituation exercises are chosen based on movements (of self or the visual environment) that provoke symptoms and the participant performs several repetitions of motions that cause mild to moderate symptoms. Balance and gait exercises are chosen based on identified impairments and limitations and are performed under challenging sensory and dynamic conditions to optimize balance. General conditioning, such as a customized graduated walking program for endurance will be included.

All participants will receive verbal instructions (in Health in Motion the text instruction is accompanied with voice over), demonstration of, and feedback on, accurate performance of the gaze stabilization/habituation HEP per group assignment. The S-VRT group will only receive these instructions and feedback at the weekly clinic visit from the supervising clinician. The D-VRT group will receive exercise instructions and demonstration via the Rock Steady app the first time using a game and as requested thereafter. The supervising clinician will evaluate the participant's ability to accurately perform the exercises at each follow-up visit (1x/week) and will provide additional training/feedback as needed for both S-VRT and D-VRT groups.

All participants will be instructed to complete the gaze stabilization/habituation exercises 2-3 times per day and the balance and gait exercises 1 time per day for 4 weeks. All participants will use a paper exercise log to record the performance of the HEP, regardless of group assignment. After completing the 4-week intervention, participants will be offered the option to continue using their current method or try the alternate method for the 3- month maintenance phase. After the 3-month maintenance phase, participants will complete the questionnaire about dizziness impact on daily activities.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age,
* diagnosis of mTBI,
* documented dizziness (total DHI score ≥ 16) and/or imbalance (total functional gait assessment score < 23/30 or < age-referenced norms)

Exclusion Criteria:

* severe neurological disease (e.g., Parkinson's disease, neuropathy),
* moderate to severe cognitive impairment (< 23/30 on the Montreal Cognitive Assessment),
* significant orthopedic issues that would impact mobility or ability to perform gaze stabilization exercises (e.g., significant cervical dysfunction or pain),
* vision impairment (best-corrected visual acuity worse than 20/40 in the better eye), and
* severe depression/anxiety (≥ 9 on the 4-item Patient health Questionnaire)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Dizziness on the Dizziness Handicap Inventory (DHI) at week four and week 12 | baseline, week 4, week 12
  The DHI is a self-report scale of the impact of dizziness on activities (Jacobson & Newman, 1990). Total scores range from 0 (no handicap) to 100 (severe handicap).

SECONDARY OUTCOMES:
Change from baseline in modified Clinical Test of Sensory Interaction and Balance (mCTSIB) at week 4 | baseline, week 4
  The mCTSIB assesses sensory integration by measuring postural stability under conditions in which visual and somatosensory feedback is altered. The test is organized into a series of four conditions of increasing difficulty. The first two conditions are performed on a firm surface with eyes open and eyes closed. The final two conditions are performed on a foam surface with eyes open and closed. The maximum duration of each trial is 30 seconds. The total score is the sum of the four conditions with a maximum total of 120 seconds.
Change from baseline in Functional Gait Assessment (FGA) at week 4 | baseline, week 4
  The FGA tests dynamic gait. The FGA is a 10-item test that incorporates more difficult gait items, e.g., head turns, narrow base of support, backwards, and with eyes closed (Wrisley et al., 2004). Total FGA scores < 23/30 indicate high fall risk and there are age-referenced norms for comparison (Walker et al., 2007).
Change from baseline in 10 Meter Walk Test (10MWT) at week 4 | baseline, week 4
  The (10MWT) will be used to assess preferred gait speed (Bohannon & Williams, 2011). Participants will walk at their normal pace on a level, 10-meter walkway. The dependent variable is preferred gait speed (m/s).
Change from baseline in Visual Analogue Scales (VAS) at week 4 | baseline, week 4
  The VAS quantifies the impact of dizziness on activities. Participants place a mark on a 10-cm horizontal line with 20% increments indicated (0-100%; Hall & Herdman, 2006). Patients indicate the percent of time that dizziness interferes with activities.
Change from baseline in Activities-specific Balance Confidence scale (ABC) at week 4 | baseline, week 4
  The ABC measures individuals' confidence that they can maintain balance in a variety of situations (Powell & Myers, 1995). The ABC was developed to assess balance confidence across a continuum of activities. An overall score is calculated and lower scores indicate worse confidence in balance ability.
Change from baseline in Disability Rating Scale (DRS) at week 4 | baseline, week 4
  The DRS is a self-report measure of the overall impact of dizziness on activities (Shepard et al., 1990). The scale involves a 6-point rating scale with 0 indicating no disability and 5 indicating long-term severe disability.
Change from baseline in modified Motion Sensitivity Test (mMST) at week 4 | baseline, week 4
  The mMST is a a measure of is a measure of motion-provoked dizziness. The test involves ten quick movements that are performed in standing and after each movement is completed, the intensity and duration of symptoms are recorded (Heusel-Gillig et al., 2022). A total score is calculated and can range from 0 to 100 with higher scores indicating greater motion sensitivity.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - James A Haley VA Hospital, Tampa, Florida
  - Duke University School of Medicine, Durham, North Carolina
  - James H Quillen VAMC, Mountain Home, Tennessee

IPD SHARING:
Plan to Share IPD: No
We will comply with VA policy regarding the dissemination of de-identified data collected from participants consenting to Federal Interagency Traumatic Brain Injury Research (FITBIR) informatics system and the FDA. We will make available descriptive data on device accuracy and effectiveness.

REFERENCES:
- [Background] Jacobson GP, Newman CW. The development of the Dizziness Handicap Inventory. Arch Otolaryngol Head Neck Surg. 1990 Apr;116(4):424-7. doi: 10.1001/archotol.1990.01870040046011. PMID 2317323
- [Background] Wrisley DM, Marchetti GF, Kuharsky DK, Whitney SL. Reliability, internal consistency, and validity of data obtained with the functional gait assessment. Phys Ther. 2004 Oct;84(10):906-18. PMID 15449976
- [Background] Walker ML, Austin AG, Banke GM, Foxx SR, Gaetano L, Gardner LA, McElhiney J, Morris K, Penn L. Reference group data for the functional gait assessment. Phys Ther. 2007 Nov;87(11):1468-77. doi: 10.2522/ptj.20060344. Epub 2007 Sep 4. PMID 17785375
- [Background] Bohannon RW, Williams Andrews A. Normal walking speed: a descriptive meta-analysis. Physiotherapy. 2011 Sep;97(3):182-9. doi: 10.1016/j.physio.2010.12.004. Epub 2011 May 11. PMID 21820535
- [Background] Hall CD, Herdman SJ. Reliability of clinical measures used to assess patients with peripheral vestibular disorders. J Neurol Phys Ther. 2006 Jun;30(2):74-81. doi: 10.1097/01.npt.0000282571.55673.ed. PMID 16796772
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Shepard NT, Telian SA, Smith-Wheelock M. Habituation and balance retraining therapy. A retrospective review. Neurol Clin. 1990 May;8(2):459-75. PMID 2359384
- [Background] Heusel-Gillig L, Santucci V, Hall CD. Development and Validation of the Modified Motion Sensitivity Test. Otol Neurotol. 2022 Sep 1;43(8):944-949. doi: 10.1097/MAO.0000000000003641. PMID 35970158